CLINICAL TRIAL: NCT01298388
Title: Assessment of the Long Term Outcome of Childhood ALL Patients Enrolled in EORTC Children's Leukemia Group Trials Between 1971 and 1998
Brief Title: Study of Long-Term Outcomes of Patients With Acute Lymphoblastic Leukemia Who Were Enrolled as Children on Clinical Trials EORTC-58741, EORTC-58831, EORTC-58832, or EORTC-58881 Between 1971 and 1998
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000695273; EORTC-58LAE; EU-21106
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Cancer Survivor; Leukemia; Long-term Effects Secondary to Cancer Therapy in Children
Keywords: long-term effects secondary to cancer therapy in children; cancer survivor; recurrent childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia; non-T, non-B childhood acute lymphoblastic leukemia; non-T, non-B, cALLa positive childhood acute lymphoblastic leukemia; non-T, non-B, cALLa negative childhood acute lymphoblastic leukemia; non-T, non-B, cALLa positive, pre-B childhood acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia in remission
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

INTERVENTIONS:
Other: medical chart review
Other: questionnaire administration
Other: study of socioeconomic and demographic variables

SUMMARY:
RATIONALE: Studying medical records and collecting questionnaires from patients who were enrolled as children in clinical trials for acute lymphoblastic leukemia may help doctors learn about long-term effects of treatment and plan the best treatment.

PURPOSE: This clinical trial is studying the long-term outcomes of patients with acute lymphoblastic leukemia who were enrolled as children on clinical trials EORTC-58741, EORTC-58831, EORTC-58832, or EORTC-58881 between 1971 and 1998.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the long-term outcomes (i.e., long-term survival, long-term disease status, occurrence of late adverse effects, occurrence of second cancers, and socioeconomic status of survivors) of patients with acute lymphoblastic leukemia previously enrolled as children on clinical trials EORTC-58741, EORTC-58831, EORTC-58832, or EORTC-58881 between the years of 1971 and 1998.

OUTLINE: Long-term outcome data are collected from the databases about clinical trials EORTC-58741, EORTC-58831, EORTC-58832, or EORTC-58881. Other data collected include the patient's vital status actualization (e.g., alive, dead or lost to follow up, date last known to be alive or date of death), medical records data, and the collection of data from patients confirmed to be alive (e.g., data related to marital status, education, work, insurance, puberty, fertility, and offspring) by questionnaire.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients with acute lymphoblastic leukemia (ALL) previously enrolled as children (less than18 years of age at diagnosis) on any of the following clinical trials between 1971 and 1998:

  * EORTC-58741
  * EORTC-58831
  * EORTC-58832
  * EORTC-58881

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3138 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Long-term survival
Disease status
Late adverse effects
Second cancers
Socioeconomic status of survivors

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Piette, Study Chair — Centre Hospitalier Regional de la Citadelle; Yves Benoit, MD — University Ghent

REFERENCES:
- [Derived] de Ville de Goyet M, Kicinski M, Suciu S, Vandecruys E, Uyttebroeck A, Ferster A, Freycon C, Plat G, Thomas C, Barbati M, Dresse MF, Paillard C, Pluchart C, Simon P, Chantrain C, Minckes O, van der Werff Ten Bosch J, Bertrand Y, Rohrlich P, Millot F, Paulus R, Benoit Y, Piette C; European Organisation for Research, Treatment of Cancer (EORTC) Children's Leukemia Group (CLG). Long-term neurotoxicity among childhood acute lymphoblastic leukaemia survivors enrolled between 1971 and 1998 in EORTC Children Leukemia Group studies. Discov Oncol. 2024 Jan 29;15(1):20. doi: 10.1007/s12672-024-00869-6. PMID 38285235
- [Derived] Rossi G, Kicinski M, Suciu S, Vandecruys E, Plat G, Uyttebroeck A, Paillard C, Barbati M, Dresse MF, Simon P, Minckes O, Pluchart C, Ferster A, Freycon C, Millot F, van der Werff Ten Bosch J, Chantrain C, Paulus R, de Rojas T, de Schaetzen G, Rohrlich P, Benoit Y, Piette C. Fertility status among long-term childhood acute lymphoblastic leukaemia survivors enrolled between 1971 and 1998 in EORTC CLG studies: results of the 58 Late Adverse Effects study. Hum Reprod. 2021 Dec 27;37(1):44-53. doi: 10.1093/humrep/deab236. PMID 34788455